CLINICAL TRIAL: NCT06779175
Title: Analysis of Single Respiratory Viral Infections Versus Co-infections in the Post-pandemic Era: Prevalence and ICU Needs in Hospitalized Adults
Brief Title: Analysis of Single Respiratory Viral Infections Versus Co-infections: Prevalence and ICU Needs in Hospitalized Adults
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Özlem Güler, Assistant Professor M.D., Kocaeli University
Other Study IDs: GOKAEK-2024/05.17 2024/140
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Tract Infections; Virus Diseases; Coinfection
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Viral respiratory infection: Symptomatic and verified viral upper respiratory tract infections in hospitalized patients
- Viral respiratory co-infection: Inpatients who are symptomatic and infected with more than one respiratory virus simultaneously

SUMMARY:
The objective of our study is to investigate the prevalence of viral respiratory infections in inpatients following the end of the pandemic. Additionally, the prevalence of patients co-infected with multiple viruses simultaneously will be assessed.

In the secondary part of the study, the development of respiratory tract infections, the need for intensive care, and mortality rates within seven days will also be evaluated, and risk factors for patients with a more severe clinical course will be statistically calculated.

DETAILED DESCRIPTION:
This study aims to determine the prevalence of viral respiratory agents in hospitalized patients post-COVID-19 and to examine the clinical course of respiratory viral co-infections, which are expected to be more severe.

This study will be conducted retrospectively at Kocaeli University Hospital between May 2023, considered the end date of the pandemic, and January 2024. Patients over 18 years of age will be included, and data will be accessed through the hospital automation system. Patients with SARS-CoV-2 PCR-positive symptoms and those expected to use molnupiravir due to the need for treatment will be considered as COVID-19. Respiratory tract agents will be detected by multiplex PCR from symptomatic inpatients. All patients with influenza will also receive oseltamivir. The distribution of viruses, the need for intensive care hospitalization, and whether they cause death within seven days, as well as the prevalence, clinical course, and risk factors of viral co-infections expected to be clinically more severe in the literature, will also be examined

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients admitted to our clinic or consulted to infectious diseases from other inpatient services.
* Patients diagnosed with upper or lower respiratory tract infections due to viral agents

Exclusion Criteria:

* Patients infected with bacterial agents will not be included in the study.
* Patients admitted from the outpatient clinic were not included in the study plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients over 18 years of age who are hospitalized, have symptoms of respiratory tract infection, and have a positive result for a respiratory tract virus detected by PCR. Patients with SARS-CoV-2 PCR-positive symptoms who require antiviral treatment will be classified as cases of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of Single and Co-infections in Respiratory Viral Infections | On 12 January 2025, the retrospective analysis of patients was started. The study is expected to be completed within 3 months.
  Objective: To determine the prevalence of single respiratory viral infections and co-infections in hospitalized adults after COVID-19 pandemic.
  Assessment Tool: Hospital automation system for patient demographic and clinical data, and multiplex PCR testing for pathogen detection.
  Unit of Measure:
  Percentage of patients with each viral infections

SECONDARY OUTCOMES:
Risk Factors and Rates of ICU Admission and Mortality in Respiratory Viral Infections | On 12 January 2025, the retrospective analysis of patients was started. The study is expected to be completed within 3 months.
  Objective: To assess the risk factors for ICU admission and seven-day mortality in patients with respiratory viral infections Assessment Tool: Patient records for ICU admission and mortality data, combined with statistical analysis to identify risk factors.
  Unit of Measure:
  Odds ratios for ICU admission and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Güler, Assist. Prof, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shan N, Zheng Z. A Case of Nosocomial Coinfection of SARS-CoV-2 and Influenza A Virus in a Hospitalized Patient with Acute Myocardial Infarction. Clin Lab. 2024 Jan 1;70(1). doi: 10.7754/Clin.Lab.2023.230735. PMID 38213216
- [Background] Kanji JN, Zelyas N, Pabbaraju K, Granger D, Wong A, Murphy SA, Buss E, MacDonald C, Berenger BM, Diggle MA, Marshall NC, Conly JM, Tipples G. Respiratory virus coinfections with severe acute respiratory coronavirus virus 2 (SARS-CoV-2) continue to be rare one year into the coronavirus disease 2019 (COVID-19) pandemic in Alberta, Canada (June 2020-May 2021). Infect Control Hosp Epidemiol. 2023 May;44(5):805-808. doi: 10.1017/ice.2021.495. Epub 2021 Dec 6. PMID 34866560
- [Background] Mochan E, Sego TJ. Mathematical Modeling of the Lethal Synergism of Coinfecting Pathogens in Respiratory Viral Infections: A Review. Microorganisms. 2023 Dec 13;11(12):2974. doi: 10.3390/microorganisms11122974. PMID 38138118